CLINICAL TRIAL: NCT02711215
Title: Patient Stratification and Treatment Response Prediction in Neuropharmacotherapy Using Hybrid Positron Emmission Tomography/Magnetic Resconance Imaging (PET/MR)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, Head of the Neuroimaging Labs, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1.6_20180316
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Multimodal Imaging; Molecular Imaging; Citalopram; Escitalopram; Mirtazapine; Dexetimide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Diagnostic Test: PET/MR [11C]DASB — 2 PET/MR scans will be performed (placebo/citalopram - double-blind randomized cross-over)
  Other Names: Hybrid imaging, Molecular imaging, SERT binding potential
Drug: Citalopram — 8mg citalopram or placebo (saline) will be applied during PET/MR measurements in a double-blind randomized cross-over design
  Other Names: Seropram
Drug: Escitalopram (Mirtazapine/Duloxetine/Venlafaxine) — After completion of imaging procedures, patients will receive treatment with escitalopram 10-20mg. In case of non-response, after 6 weeks, treatment will be switched to either Mirtazapine, Duloxetine or Venlafaxine
  Other Names: Cipralex
Drug: Placebo — 8mg citalopram or placebo (saline) will be applied during PET/MR measurements in a double-blind randomized cross-over design
  Other Names: Saline, NaCL

SUMMARY:
Selective serotonin reuptake inhibitors (SSRIs) raise serotonin (5-HT) in the synaptic cleft and are the current first line of pharmacological antidepressive treatment. Yet, there is a missing link between this first molecular step in their mechanism of action and observed clinical improvement. We have determined to establish a framework combining genuine molecular and functional imaging, i.e. hybrid pharmaco-PET/MR imaging, of the human serotonergic system in order to predict antidepressant treatment response.

Objectives:

1. To predict antidepressant treatment response from data obtained using hybrid PET/MR with acute pharmacological challenge.
2. To discriminate healthy from depressed subjects using this paradigm.
3. To establish models connecting regional changes in occupancy of serotonin transporters (5-HTT) following citalopram infusion, with changes in brain activation and connectivity of major resting-state hub networks.

Design: Randomized, double-blind, placebo-controlled, cross-over mono-center study.

Materials and methods:

40 major depressed (MDD) and 40 healthy subjects will undergo 2 PET/MR scans on a 3T SIEMENS mMR Biograph scanner: 1. challenge with citalopram 8mg 2. placebo (saline). After structural imaging, functional MRI will be continuously acquired. [11C]DASB will be applied using a bolus + constant infusion paradigm to probe 5-HTT binding potentials and monitor 5-HTT occupancy with drug challenge, applied after 70min, in a single session. Scanning will be terminated 80min after challenge. MDD patients will receive subsequent escitalopram treatment with repeated evaluation of response for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* General health based on medical history, physical examination and structured clinical interview for DSM-IV (SCID)
* HAM-D≥18 (patients)
* Willingness and competence to sign the informed consent form
* Age 18 to 55 years

Exclusion Criteria:

* Any medical, psychiatric or neurological illness (other than MDD)
* Current or former psychopharmacological treatment
* Current or former substance abuse
* Pregnancy
* Any implant or stainless steel graft or any other contraindications for MRI
* Failure to comply with the study protocol or to follow the instructions of the investigating team
* Participation in studies involving radiation exposure in the past 10 years.
* Body mass index <17 or >30

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-05; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale (HDRS) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Zadka L, Eggerstorfer B, Buzalewicz I, Vraka C, Rusak A, Godbersen GM, Opalinska A, Unterholzner J, Ulatowska-Jarza A, Philippe C, Haczkiewicz-Lesniak K, Silberbauer LR, Murgas M, Nics L, Hahn A, Hacker M, Gomulkiewicz A, Rujescu D, Podhorska-Okolow M, Lanzenberger R, Gryglewski G. Phenotyping extracellular vesicles and their serotonin transporter cargo in major depressive disorder. J Affect Disord. 2025 Nov 15;389:119740. doi: 10.1016/j.jad.2025.119740. Epub 2025 Jun 21. PMID 40550277
- [Derived] Seiger R, Gryglewski G, Klobl M, Kautzky A, Godbersen GM, Rischka L, Vanicek T, Hienert M, Unterholzner J, Silberbauer LR, Michenthaler P, Handschuh P, Hahn A, Kasper S, Lanzenberger R. The Influence of Acute SSRI Administration on White Matter Microstructure in Patients Suffering From Major Depressive Disorder and Healthy Controls. Int J Neuropsychopharmacol. 2021 Jul 23;24(7):542-550. doi: 10.1093/ijnp/pyab008. PMID 33667309